CLINICAL TRIAL: NCT04724356
Title: Effect of Exercise Mode on Physical Function and Quality of Life in Breast Cancer-Related Lymphedema: A Randomized Controlled Trial
Brief Title: Effect of Exercise Mode in Breast Cancer-Related Lymphedema
Acronym: Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, Department of Physical Therapy, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah., Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2449PT
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer Lymphedema; Quality of Life
MeSH Terms: conditions — Breast Cancer Lymphedema | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): The Kinect based rehabilitation group received virtual reality therapy using Xbox Kinect-based games, in addition to complex decongestive physiotherapy. The intervention was led once per day, five days a week, over 8 weeks. All participants wearing multilayer bandage or compression stocking during training to avoid exacerbation of the lymphedema in the affected limb.
  Interventions: Other: Virtual Reality
- Resistance exercise Group (Experimental): The resistance exercise group received resistance training, in addition to complex decongestive physiotherapy. The intervention was led once per day, five days a week, over 8 weeks. All participants wearing multilayer bandage or compression stocking during training to avoid exacerbation of the lymphedema in the affected limb.
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Virtual Reality — Intervention was led once per day, five days a week, over 8 weeks.
  Other Names: complex decongestive physiotherapy
  Arms: Virtual Reality Group
Other: Resistance Exercise — Intervention was led once per day, five days a week, over 8 weeks.
  Other Names: complex decongestive physiotherapy
  Arms: Resistance exercise Group

SUMMARY:
Gaining a greater understanding of how each exercise mode affects lymphedema, as well as other health-related outcomes will improve exercise prescription guidelines relevant to this specific lymphedema. Therefore, the purpose of this work was to compare the effects of Xbox kinect rehabilitation and resistance exercises on limb volume, symptoms severity, physical function, and quality of life in women with Breast cancer-related lymphedema.

DETAILED DESCRIPTION:
Breast cancer-related lymphedema is a common and debilitating side effect of cancer treatment. This study compared the effect of Xbox kinect rehabilitation and resistance exercises on breast cancer-related lymphedema volume and severity, as well as participant's physical function and quality of life. Women diagnosed with unilateral breast cancer related lymphedema were randomly divided into two groups: the kinect based rehabilitation group KBRG and resistance exercise group REG. woman in The KBRG received virtual reality therapy using Xbox Kinect-based games, the REG received resistance training in addition both groups received complex decongestive physiotherapy. The intervention was five sessions per week for 8 weeks. The outcome measures included limb volume, symptoms severity, physical function (muscle strength and range of motion) and quality of life. All these outcomes were assessed at pretreatment (baseline) and after the end of treatment at week eight (W8).

ELIGIBILITY:
Inclusion Criteria:

* Age more than 30.
* Histological diagnosis of breast cancer at least 1 year prior to the study.
* Clinical diagnosis of unilateral Breast cancer-related lymphedema and obtained medical clearance from their medical oncologists or surgeons.
* Clinical diagnosis of lymphedema was defined as having at least a 5 % inter-limb discrepancy in volume or circumference.

Exclusion Criteria:

* Unstable lymphedema, receiving intensive therapy within the previous 3 months.
* A musculoskeletal, cardiovascular and/or neurological disorder that could inhibit them from exercising.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer-Related Lymphedema
Enrollment: 52 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Limb volume measurement | at baseline
  assessed by circumference measurements using a non-elastic tape. Measures started just distal to the metacarpal-phalangeal joints and were taken at 4-cm intervals up the arm until the base of the axilla.
Limb volume measurement | after 8 weeks
  assessed by circumference measurements using a non-elastic tape. Measures started just distal to the metacarpal-phalangeal joints and were taken at 4-cm intervals up the arm until the base of the axilla.
Limb volume measurement | after 12 weeks
  assessed by circumference measurements using a non-elastic tape. Measures started just distal to the metacarpal-phalangeal joints and were taken at 4-cm intervals up the arm until the base of the axilla.
Health-related quality of life, Medical Outcomes Study short-form (SF-36) | at baseline
  assessed using the Medical Outcomes Study short-form (SF-36). Outcomes of physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role emotional and mental health domains were reported as norm-based scores.
Health-related quality of life, Medical Outcomes Study short-form (SF-36) | after 8 weeks
  assessed using the Medical Outcomes Study short-form (SF-36). Outcomes of physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role emotional and mental health domains were reported as norm-based scores.
Health-related quality of life, Medical Outcomes Study short-form (SF-36) | after 12 weeks
  assessed using the Medical Outcomes Study short-form (SF-36). Outcomes of physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role emotional and mental health domains were reported as norm-based scores.

SECONDARY OUTCOMES:
Shoulder range of motion | at baseline
  Active flexion and abduction of the shoulder were assessed with the elbow extended in the supine position. External rotation was measured while the shoulder was adducted and in neutral position with the forearm in neutral supination and pronation while sitting on a chair.
Shoulder range of motion | after 8 weeks
  Active flexion and abduction of the shoulder were assessed with the elbow extended in the supine position. External rotation was measured while the shoulder was adducted and in neutral position with the forearm in neutral supination and pronation while sitting on a chair.
Shoulder range of motion | after 12 weeks
  Active flexion and abduction of the shoulder were assessed with the elbow extended in the supine position. External rotation was measured while the shoulder was adducted and in neutral position with the forearm in neutral supination and pronation while sitting on a chair.
Visual analogue scale | at baseline
  used to quantify the severity of perceived pain, heaviness, and tightness. Participants rated their symptom severity from no pain/no discomfort (score = 0) to very severe pain/worst imaginable discomfort (score = 10)
Visual analogue scale | after 8 weeks
  used to quantify the severity of perceived pain, heaviness, and tightness. Participants rated their symptom severity from no pain/no discomfort (score = 0) to very severe pain/worst imaginable discomfort (score = 10)
Visual analogue scale | after 12 weeks
  used to quantify the severity of perceived pain, heaviness, and tightness. Participants rated their symptom severity from no pain/no discomfort (score = 0) to very severe pain/worst imaginable discomfort (score = 10)
Muscle strength | at baseline
  The affected upper extremity flexion, abduction, and external rotation muscle strength were measured during maximal voluntary isometric muscle contraction with the J Tech Commender Muscle Tester (Salt Lake City, Utah, USA) handheld dynamometer according to reported positions.
Muscle strength | after 8 weeks
  The affected upper extremity flexion, abduction, and external rotation muscle strength were measured during maximal voluntary isometric muscle contraction with the J Tech Commender Muscle Tester (Salt Lake City, Utah, USA) handheld dynamometer according to reported positions.
Muscle strength | after 12 weeks
  The affected upper extremity flexion, abduction, and external rotation muscle strength were measured during maximal voluntary isometric muscle contraction with the J Tech Commender Muscle Tester (Salt Lake City, Utah, USA) handheld dynamometer according to reported positions.

CONTACTS AND LOCATIONS:
Overall Officials: Maged Basha, PhD, Principal Investigator — College of medical rehabilitation, Qassim University; Fatma Alzahraa Kamel, PhD, Study Director — Cairo University
Locations (1):
- Shorook Physical Therapy Centers, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Vicini F, Shah C, Arthur D. The Increasing Role of Lymphedema Screening, Diagnosis and Management as Part of Evidence-Based Guidelines for Breast Cancer Care. Breast J. 2016 May;22(3):358-9. doi: 10.1111/tbj.12586. Epub 2016 Feb 29. No abstract available. PMID 26929240
- [Background] Morgan PA, Franks PJ, Moffatt CJ. Health-related quality of life with lymphoedema: a review of the literature. Int Wound J. 2005 Mar;2(1):47-62. doi: 10.1111/j.1742-4801.2005.00066.x. PMID 16722853
- [Result] Aguilar-Lazcano CA, Rechy-Ramirez EJ, Hu H, Rios-Figueroa HV, Marin-Hernandez A. Interaction Modalities Used on Serious Games for Upper Limb Rehabilitation: A Systematic Review. Games Health J. 2019 Oct;8(5):313-325. doi: 10.1089/g4h.2018.0129. Epub 2019 Jul 9. PMID 31287734
- [Derived] Basha MA, Aboelnour NH, Alsharidah AS, Kamel FH. Effect of exercise mode on physical function and quality of life in breast cancer-related lymphedema: a randomized trial. Support Care Cancer. 2022 Mar;30(3):2101-2110. doi: 10.1007/s00520-021-06559-1. Epub 2021 Oct 20. PMID 34669036